CLINICAL TRIAL: NCT02873195
Title: BACCI: A Phase II Randomized, Double-Blind, Placebo-Controlled Study of Capecitabine Bevacizumab Plus Atezolizumab Versus Capecitabine Bevacizumab Plus Placebo in Patients With Refractory Metastatic Colorectal Cancer
Brief Title: Capecitabine and Bevacizumab With or Without Atezolizumab in Treating Patients With Refractory Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RU021416I; NCI-2016-01263 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RU021416I (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Colorectal Carcinoma; Recurrent Colorectal Carcinoma; Refractory Colorectal Carcinoma; Stage IV Colorectal Cancer AJCC v7; Stage IVA Colorectal Cancer AJCC v7; Stage IVB Colorectal Cancer AJCC v7
MeSH Terms: conditions — Colorectal Neoplasms | interventions — atezolizumab; Bevacizumab; Immunoglobulin G; Disulfides; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (atezolizumab, bevacizumab, capecitabine) (Experimental): Patients receive atezolizumab IV over 30-60 minutes on day 1, bevacizumab IV over 30-90 minutes on day 1, and capecitabine PO BID on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Biological: Bevacizumab; Drug: Capecitabine; Other: Laboratory Biomarker Analysis
- Arm II (placebo, bevacizumab, capecitabine) (Active Comparator): Patients receive placebo IV over 30-60 minutes on day 1, bevacizumab IV over 30-90 minutes on day 1, and capecitabine PO BID on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Capecitabine; Other: Laboratory Biomarker Analysis; Other: Placebo

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
  Arms: Arm I (atezolizumab, bevacizumab, capecitabine)
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo — Given IV
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo, bevacizumab, capecitabine)

SUMMARY:
This randomized phase II trial studies how well capecitabine and bevacizumab with or without atezolizumab work in treating patients with colorectal cancer that is not responding to treatment and has spread to other places. Immunotherapy with monoclonal antibodies, such as atezolizumab and bevacizumab, may help the body?s immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving atezolizumab with capecitabine and bevacizumab may be a better way in treating colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the efficacy of capecitabine/bevacizumab + atezolizumab, as compared with capecitabine/bevacizumab + placebo in refractory metastatic colorectal cancer (mCRC) as measured by progression-free survival (defined as the time of randomization to the first occurrence of progression based on Response Evaluation Criteria in Solid Tumors version 1.1, clinical progression, or death from any cause on study as determined by the investigator).

SECONDARY OBJECTIVES:

I. To estimate the efficacy of capecitabine/bevacizumab + atezolizumab, as compared with capecitabine/bevacizumab + placebo in refractory mCRC as measured by objective response rate (defined as partial response plus complete response) as determined by the investigator using Response Evaluation Criteria in Solid Tumors version 1.1 and immune-related response criteria (irRC).

II. To estimate the efficacy of capecitabine/bevacizumab + atezolizumab as compared with capecitabine/bevacizumab + placebo in refractory mCRC as measured by overall survival (defined as death from any cause from the time of randomization until study completion).

III. To evaluate the safety and tolerability of atezolizumab in combination with bevacizumab and capecitabine in refractory mCRC as measured by the serious adverse events and adverse events >= grade 3 according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.

CORRELATIVE OBJECTIVE:

I. To explore any correlation between tissue and blood based biomarkers and clinical outcomes.

OUTLINE: Patients are randomized 2:1 to Arm I:Arm II.

ARM I (ATEZOLIZUMAB, BEVACIZUMAB, CAPECITABINE): Patients receive atezolizumab intravenously (IV) over 30-60 minutes on day 1, bevacizumab IV over 30-90 minutes on day 1, and capecitabine orally (PO) twice daily (BID) on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM II (PLACEBO, BEVACIZUMAB, CAPECITABINE): Patients receive placebo IV over 30-60 minutes on day 1, bevacizumab IV over 30-90 minutes on day 1, and capecitabine PO BID on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 3 months until progressive disease, then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal cancer that is either clinically or histologically proven to be metastatic and has progressed on regimens containing a fluoropyrimidine (e.g., 5-fluorouracil or capecitabine), oxaliplatin, irinotecan, bevacizumab and an anti-EGFR antibody (if tumor is RAS wild-type), or where the treatment was not tolerated or contraindicated
* Measurable disease; Note: previously irradiated sites can be included if there is documented disease progression in that site
* Capecitabine and bevacizumab considered appropriate treatment for the patient
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Absolute neutrophil count >= 1,500/uL (obtained =< 7 days prior to randomization)
* Platelets >= 100,000/uL (obtained =< 7 days prior to randomization)
* Total bilirubin =< 1.5 X upper limit of normal (ULN) (obtained =< 7 days prior to randomization); patients with known Gilbert?s syndrome who have serum bilirubin =< 3 X ULN may enroll
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 1.5 X ULN; < 3 X ULN if known hepatic metastases (obtained =< 7 days prior to randomization)
* Hemoglobin >= 9 g/dL continuation of erythropoietin products is permitted (obtained =< 7 days prior to randomization); hemoglobin must be stable >= 9 g/dL >= 14 days without blood transfusion to maintain hemoglobin level
* Calculated creatinine clearance must be >= 50 ml/min using the Cockcroft-Gault formula or a 24 hour urine (obtained =< 7 days prior to randomization)
* The following laboratory values obtained =< 14 days prior to randomization

  * Prothrombin time (PT)/partial thromboplastin time (PTT)/international normalized ratio (INR) =< 1.5 X ULN if not anticoagulated; within local institutional guidelines per local physician if anticoagulated
* Negative pregnancy test done =< 7 days prior to randomization, for women of childbearing potential only
* Provide informed written consent
* Willingness to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willingness to provide tissue and blood samples for correlative research purposes
* Life expectancy of >= 3 months

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
  * Women of child-bearing potential must agree to use two forms of adequate contraception from time of initial consent, for the duration of study participation, and for >= 6 months after the last dose of study drug; medically acceptable contraceptives include: (1) surgical sterilization (such as a tubal ligation or hysterectomy), (2) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), (3) barrier methods (such as a condom or diaphragm) used with a spermicide, or (4) an intrauterine device (IUD); contraceptive measures such as Plan B, sold for emergency use after unprotected sex, are not acceptable methods for routine use; postmenopausal woman must have been amenorrheic for at least 2 years to be considered of non-childbearing potential; sexually active men must use at least one form of adequate contraception from time of initial consent, for the duration of study participation, and for >= 6 months after the last dose of study drug
* Chemotherapy, biologic anti-cancer therapy, or central field radiation therapy =< 28 days prior to randomization; Note: local or stereotactic radiation =< 14 days prior to randomization
* Any investigational agent =< 28 days or 5 half-lives prior to randomization (whichever is longer)
* Prior treatment with atezolizumab or another PD-L1/PD-1 therapy
* History of allergic reactions attributed to therapeutic antibodies; Note: patients with reactions to chimeric antibodies may be permitted on a case by case basis with approval by study chair by contacting the data manager
* Known untreated central nervous system (CNS) metastases; Note: patients with radiated or resected lesions are permitted, provided the lesions are fully treated and inactive, patients are asymptomatic, and no steroids have been administered for this purpose =< 30 days prior to randomization
* Inadequately controlled hypertension (defined as average systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg)
* History of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) grade II or greater congestive heart failure
* History of myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or surgery =< 12 months prior to randomization
* Active coronary heart disease evidenced as angina or requiring medications to prevent angina
* History of stroke or transient ischemic attack, or other arterial thrombosis =< 12 months prior to randomization
* Symptomatic peripheral vascular disease
* Any other significant vascular disease (e.g., aortic aneurysm, aortic dissection, or carotid stenosis that requires medical or surgical intervention, including angioplasty or stenting)
* Any previous National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade 4 venous thromboembolism
* Clinically-significant evidence of bleeding diathesis or coagulopathy as so judged by the treating physician
* History of active gastrointestinal (GI) bleeding or other major bleeding =< 12 months prior to randomization; Note: patients who do not have resolution of the predisposing risk factor (e.g., resection of a bleeding tumor, treatment and endoscopic documentation of a resolved ulcer) will also be excluded
* Major surgical procedure, open biopsy, or significant traumatic injury =< 56 days prior to randomization
* Anticipation of need for major surgical procedure =< 6 months after randomization
* Minor surgical procedure =< 7 days prior to randomization; exception: insertion of an indwelling catheter or percutaneous needle biopsy =< 48 hours prior to randomization
* History of intra-abdominal abscess =< 6 months prior to randomization; Note: if the affected area was surgically resected, and there is no further risk to the area, patients may enroll
* History of abdominal or other significant fistula, gastrointestinal or other organ perforation; Note: if the affected area was surgically resected, and there is no further risk to the area, patients may enroll
* Serious, non-healing wound, ulcer, or bone fracture as so judged by the treating physician
* Known proteinuria defined by >= 2+ protein by urinalysis (UA) or >= 1 gram protein by 24 hour urine collection; Note: Subjects that are >= 2+ or greater on dipstick but < 1 g protein on 24 hour urine ARE eligible to participate
* Intolerance to bevacizumab defined as any NCI CTCAE grade 3 or grade 4 toxicity attributed to this agent that required discontinuation of bevacizumab (e.g., arterial thromboembolism [ATE], perforation, wound healing difficulty, proteinuria, reversible posterior leukoencephalopathy syndrome [RPLS]); Note: patients with prior grade 3 bevacizumab-related hypertension may be permitted if hypertension was manageable with standard oral antihypertensives as so judged by the treating physician
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Impairment of GI function or GI disease that may significantly alter capecitabine drug absorption
* Active inflammatory bowel disease
* History of diverticulitis, chronic ulcerative lower GI disease such as Crohn?s disease or ulcerative colitis, or other symptomatic lower GI conditions that might predispose to perforations
* History of autoimmune disease including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener?s granulomatosis, Sjogren?s syndrome, Bell?s palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis; Note: patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study
* Active current infection or history of recurrent bacterial, viral, fungal, mycobacterial or other infections, including but not limited to tuberculosis and atypical mycobacterial disease, hepatitis B and C, herpes zoster, and human immunodeficiency virus (HIV), but excluding fungal infections of nail beds
* Vaccination with a live or attenuated vaccine =< 28 days prior to randomization; Note: other types of vaccines, including inactivated/killed, toxoid (inactivated toxoid), and subunit/conjugate are all permitted at any time
* Any reversible treatment-related toxicity that has not resolved to NCI CTCAE grade =< 1 except neuropathy
* Other concurrent severe and/or uncontrolled medical disease, psychiatric illness, or social situation, which could compromise safety of treatment as so judged by the treating physician; Note: this includes but is not limited to: severely impaired lung function, uncontrolled diabetes (history of consistent blood glucose readings above 300 mg/dL or less than 50 mg/dL), severe infection, severe malnutrition, ventricular arrhythmias, known active vasculitis of any cause, tumor invasion of any major blood vessel, chronic liver or renal disease, and active upper GI tract ulceration
* Unwilling to or unable to comply with the protocol
* Current or recent (=< 10 days prior to randomization) use of aspirin (> 325 mg/day), or clopidogrel (> 75 mg/day)
* Current or recent (=< 10 days prior to randomization) use of therapeutic oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes, unless the patient has been on a stable dose of anticoagulants for at least 2 weeks at the time of randomization; Note: the use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or activated partial thromboplastin time (aPTT) is within therapeutic limits (according to the medical standard of the institution) and the patient has been on a stable dose of anticoagulants >= 14 days at the time of randomization; prophylactic use of anticoagulants is allowed
* History or recent diagnosis of demyelinating disease
* History of other carcinoma =< 3 years; exception: if risk of recurrence is known to be under 5% at time of randomization
* Current or recent (=< 90 days prior to randomization) endoluminal stent in the stomach, bowel, colon or rectum
* Colonoscopy, sigmoidoscopy, or proctoscopy =< 7 days prior to randomization
* Current or recent (=< 28 days prior to randomization) use of sorivudine, brivudine, and St. John?s wort
* Primary or secondary immunodeficiency (history of or currently active) unless related to primary disease under investigation
* Prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) =< 14 days prior to randomization; exception: patients who have received acute, low-dose, systemic immunosuppressant medications (e.g. a one-time dose of dexamethasone for nausea) are eligible; the use of inhaled corticosteroids and mineral-corticoids (e.g. fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niharika Mettu, Principal Investigator — Academic and Community Cancer Research United
Locations (10):
- United States (10):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Mettu NB, Ou FS, Zemla TJ, Halfdanarson TR, Lenz HJ, Breakstone RA, Boland PM, Crysler OV, Wu C, Nixon AB, Bolch E, Niedzwiecki D, Elsing A, Hurwitz HI, Fakih MG, Bekaii-Saab T. Assessment of Capecitabine and Bevacizumab With or Without Atezolizumab for the Treatment of Refractory Metastatic Colorectal Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2022 Feb 1;5(2):e2149040. doi: 10.1001/jamanetworkopen.2021.49040. PMID 35179586

RESULTS

PARTICIPANT FLOW:
Groups:
- Atezolizumab, Bevacizumab, Capecitabine: Patients receive 1200 mg atezolizumab IV over 30-60 minutes on day 1, 7.5 mg/kg bevacizumab IV over 30-90 minutes on day 1, and 850 or 1000 mg/m^2 capecitabine PO BID on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Placebo, Bevacizumab, Capecitabine: Patients receive 1200 mg placebo IV over 30-60 minutes on day 1, 7.5 mg/kg bevacizumab IV over 30-90 minutes on day 1, and 850 or 1000 mg/m^2 capecitabine PO BID on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Atezolizumab, Bevacizumab, Capecitabine | Placebo, Bevacizumab, Capecitabine
Started | 87 | 46
Never Began Treatment (Cancel) (Participants who never began treatment are not evaluable for adverse events.) | 1 | 0
Completed (Modified Intent-to-treat (ITT) population) | 82 | 46
Not Completed | 5 | 0
Not completed — Ineligible | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atezolizumab, Bevacizumab, Capecitabine | Placebo, Bevacizumab, Capecitabine | Total
Number analyzed (Participants) | 82 | 46 | 128
Age, Continuous [Median (Full Range); unit: years] | 59 [39 to 83] | 56 [39 to 80] | 58 [39 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 16 | 51
  Male | 47 | 30 | 77
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 7 | 8 | 15
  White | 66 | 36 | 102
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 39 | 21 | 60
    1 | 43 | 25 | 68

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. The primary comparisons will be superiority of the active treatment for PFS of atezolizumab versus placebo. PFS will be compared between treatment arms using the un-stratified log-rank test at one-sided level of 0.10 and the p-value will be used for decision making. The hazard ratio (HR) for PFS will be estimated using a Cox proportional hazards model and the 95% confidence interval (CI) for the HR will be provided. Kaplan-Meier methodology will be used to estimate the median PFS for each treatment arm, and Kaplan-Meier curves will be produced. Progression is defined as any new lesion or increase by ≥20% of previously involved sites from nadir based on RECIST criteria.
Time Frame: From randomization to first documentation of disease progression by RECIST v1.1, or death from any cause, assessed up to 20 months
Population: Modified Intent-to-treat (ITT) population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab, Bevacizumab, Capecitabine | Placebo, Bevacizumab, Capecitabine
Number analyzed (Participants) | 82 | 46
months | 4.37 [4.07 to 6.41] | 3.32 [2.14 to 6.21]
Statistical Analysis 1: Comparison: Atezolizumab, Bevacizumab, Capecitabine vs Placebo, Bevacizumab, Capecitabine; Test type: Superiority; p = 0.051, Log Rank; Hazard Ratio (HR) = 0.725, 95% CI 2-sided [0.491 to 1.07]

2. Secondary Outcome: Overall Survival (OS)
Description: The distribution of survival time will be estimated using the method of Kaplan-Meier. OS will be compared between treatment arms using the unstratified log-rank test. OS medians, survival rates and HR will be estimated along with 95% confidence intervals.
Time Frame: From randomization to death due to any cause, assessed up to 20 months
Population: Modified Intent-to-treat (ITT) population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab, Bevacizumab, Capecitabine | Placebo, Bevacizumab, Capecitabine
Number analyzed (Participants) | 82 | 46
months | 10.55 [8.21 to NA] — The 95% confidence interval upper limit was not reached (below the level of detection). | 10.61 [8.80 to NA] — The 95% confidence interval upper limit was not reached (below the level of detection).
Statistical Analysis 1: Comparison: Atezolizumab, Bevacizumab, Capecitabine vs Placebo, Bevacizumab, Capecitabine; Test type: Superiority; p = 0.40, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.56 to 1.56]

3. Secondary Outcome: Objective Response Rate
Description: The objective response rate is defined as the percentage of participants who achieve a partial response or compete response as assessed (partial response [PR] or complete response [CR] per RECIST v1.1) during treatment with study therapy. Rates of response will be compared across arms using a fisher's exact test for proportion. Point estimates will be generated for objective response rates within each arm along with 95% binomial confidence intervals. Complete response (CR): Disappearance of all evidence of disease, Partial response (PR): Regression of measurable disease and no new sites
Time Frame: Up to 20 months
Population: Modified Intent-to-treat (ITT) population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab, Bevacizumab, Capecitabine | Placebo, Bevacizumab, Capecitabine
Number analyzed (Participants) | 82 | 46
percentage of participants | 8.54 [3.5 to 16.8] | 4.35 [0.53 to 14.84]
Statistical Analysis 1: Comparison: Atezolizumab, Bevacizumab, Capecitabine vs Placebo, Bevacizumab, Capecitabine; Test type: Superiority; p = 0.4876, Fisher Exact

4. Secondary Outcome: The Number of Participants Who Experienced at Least One Grade 3 or Higher Adverse Event Deemed at Least Possibly Related to Treatment (Toxicity)
Description: The number of participants who experienced at least one grade 3 or higher adverse event deemed at least possibly related to treatment (toxicity) is reported below. Graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Toxicities will be evaluated via the ordinal CTCAE standard toxicity grading.
Time Frame: Up to 20 months
Population: Participants who started treatment and are evaluable for adverse events are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab, Bevacizumab, Capecitabine | Placebo, Bevacizumab, Capecitabine
Number analyzed (Participants) | 81 | 46
Participants | 27 | 11

ADVERSE EVENTS:
Time Frame: Up to 20 months
Description: Participants who started treatment and were assessed for adverse events are summarized below.
Arm/Group | Atezolizumab, Bevacizumab, Capecitabine | Placebo, Bevacizumab, Capecitabine
All-Cause Mortality (participants affected / at risk) | 45/82 | 23/46
Serious Adverse Events (participants affected / at risk) | 36/81 | 12/46
Other Adverse Events (participants affected / at risk) | 77/81 | 42/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab, Bevacizumab, Capecitabine (N=81) | Placebo, Bevacizumab, Capecitabine (N=46)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Death NOS (General disorders) | 7 (8) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 4 (4) | 0 (0)
Flu like symptoms (General disorders) | 2 (2) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Sudden death NOS (General disorders) | 1 (1) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Papulopustular rash (Infections and infestations) | 1 (1) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 6 (11) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab, Bevacizumab, Capecitabine (N=81) | Placebo, Bevacizumab, Capecitabine (N=46)
Anemia (Blood and lymphatic system disorders) | 12 (36) | 7 (12)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 3 (9) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 21 (49) | 7 (18)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 3 (9) | 1 (1)
Constipation (Gastrointestinal disorders) | 17 (31) | 5 (5)
Dental caries (Gastrointestinal disorders) | 1 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 47 (117) | 14 (45)
Dry mouth (Gastrointestinal disorders) | 4 (15) | 1 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (11) | 1 (1)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 2 (3) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 14 (28) | 4 (7)
Nausea (Gastrointestinal disorders) | 44 (123) | 20 (42)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 26 (41) | 13 (24)
Chills (General disorders) | 3 (5) | 1 (1)
Edema limbs (General disorders) | 7 (21) | 2 (14)
Fatigue (General disorders) | 72 (369) | 34 (161)
Fever (General disorders) | 8 (11) | 1 (1)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 3 (6)
Pain (General disorders) | 5 (7) | 2 (3)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 2 (2) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 2 (2) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Pleural infection (Infections and infestations) | 0 (0) | 1 (2)
Rhinitis infective (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 2 (7) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (8) | 2 (2)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (5) | 2 (2)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (4)
Alkaline phosphatase increased (Investigations) | 3 (6) | 5 (9)
Aspartate aminotransferase increased (Investigations) | 4 (6) | 4 (4)
Blood bilirubin increased (Investigations) | 12 (24) | 7 (14)
CPK increased (Investigations) | 0 (0) | 1 (5)
Creatinine increased (Investigations) | 6 (8) | 1 (1)
INR increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 5 (33) | 4 (9)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (3) | 1 (2)
Platelet count decreased (Investigations) | 11 (38) | 7 (19)
Serum amylase increased (Investigations) | 2 (7) | 0 (0)
Weight loss (Investigations) | 3 (12) | 2 (3)
White blood cell decreased (Investigations) | 1 (2) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 19 (33) | 9 (14)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (4) | 6 (15)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (16) | 1 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (8) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 6 (7) | 4 (8)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (10) | 3 (12)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (9) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (9) | 6 (10)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 2 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (11) | 3 (5)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 11 (69) | 10 (28)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (6) | 4 (9)
Acute kidney injury (Renal and urinary disorders) | 2 (4) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (7) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 10 (24) | 8 (21)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (2) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (21) | 4 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (11) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (6)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (8) | 3 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (21) | 4 (8)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 33 (89) | 16 (57)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (4)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 9 (22) | 2 (13)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (13) | 2 (2)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 20 (66) | 14 (59)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Thromboembolic event (Vascular disorders) | 3 (8) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT02873195/Prot_SAP_000.pdf